CLINICAL TRIAL: NCT04514380
Title: Ultrasound Assessment of Gastric Volume in Elderly Patients Undergoing Total Knee Arthroplasty After Drinking Carbohydrate-containing Fluids: A Prospective Observational Non-randomized Comparative Study
Brief Title: Effect of Drinking Carbohydrate-containing Fluids on Gastric Residual Volume in Elderly Patients
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2008/633-301
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group C: Patients drank carbohydrate fluid 2 hours prior to surgery according to the routine fasting protocol by surgeon A.
  Interventions: Other: Carbohydrate fluid
- Group N: Patients did not drink carbohydrate fluid 2 hours prior to surgery according to the routine fasting protocol by surgeon B.
  Interventions: Other: Non-carbohydrate fluid

INTERVENTIONS:
Other: Carbohydrate fluid — 400 mL carbohydrate fluid
  Groups: Group C
Other: Non-carbohydrate fluid — 0 mL carbohydrate fluid
  Groups: Group N

SUMMARY:
In the past, some guidelines advised no oral intake for at least 8 hours before any surgery. However, research has shown risks associated with excessive fasting, such as postoperative insulin resistance, and advantages in shorter fasting protocols, such as reduced postoperative nausea and vomiting.

The perioperative fasting guidelines of the European Society of Anaesthesiology focus on preoperative carbohydrates. They hold that it is safe for patients to drink carbohydrate-rich fluids up to 2 hours before elective surgery and that drinking carbohydrate-rich fluids improves subjective well-being, reduces thirst and hunger, and reduces postoperative insulin resistance at an evidence level of 1++. Nevertheless, data on drinking carbohydrate fluids before surgery in elderly patients are limited.

In our institution, there are two clinical pathways for total knee arthroplasty according to the surgeons. One difference is whether carbohydrate fluids drink or not before surgery. The purpose of this study, therefore, is to assess gastric volume in fasted elderly patients using ultrasound after they drank carbohydrate fluids 2 hours before surgery and to compare with matched patients using age, body mass index, and comorbidity, who did not drink carbohydrate fluids before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty
* Age: 65~85 yeas
* ASA 1~3

Exclusion Criteria:

* Age < 65 years
* ASA >= 4
* Diabetes mellitus
* Chronic kidney disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Gastric volume | During the gastric volume measuring at preoperative holding area/ an average of 30 minutes
  Gastric volume measured before induction of spinal anesthesia using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Seok Na, MD., PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Shin HJ, Koo BW, Lim D, Na HS. Ultrasound assessment of gastric volume in older adults after drinking carbohydrate-containing fluids: a prospective, nonrandomized, and noninferiority comparative study. Can J Anaesth. 2022 Sep;69(9):1160-1166. doi: 10.1007/s12630-022-02262-9. Epub 2022 Apr 21. PMID 35449247